CLINICAL TRIAL: NCT06735183
Title: Pre-Anesthesia Visit: Analysis of Coverage Rate of Pre-Anesthesia Visit Content by Anesthesiology Residents, and Surgical Patients' Understanding of Pre-Anesthesia Visit Information
Brief Title: Pre-Anesthesia Visit: Analysis of Coverage Rate of Visit Content and Surgical Patients' Understanding of Information
Acronym: Pre-Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Anshi Wu (Other)
Responsible Party: Sponsor-Investigator, Anshi Wu, Administrative Director of Anesthesiology, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: PAV20241212; Pre-Anesthesia Visit (Registry Identifier: PAV20241212)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: To Assess the Coverage of Anesthesiology Residents' Explanations of the Content of the Visit; Patients' Understanding of the Content of the Anesthesia Approach Through the Physician's Explanations
Keywords: preoperative anesthesia visit; understanding of the content of the anesthesia approach

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Group: To investigate patients' understanding of the content of the anesthesia visit after listening to the visit. A questionnaire was used to collect data.
  The questionnaire included the contents of the visit that the patients could recall, their understanding of the physician's explanation, their concerns, and their suggestions for improving the preoperative visit.

SUMMARY:
The aim of this study was to systematically assess the coverage of anesthesiology residents' explanations of the content of the visit during the preoperative anesthesia visit and the patients' understanding of the content of the anesthesia approach through the physician's explanations.

DETAILED DESCRIPTION:
Physician Component:

In order to minimize the change of the interview content due to third-party supervision, the collected data were analyzed in the form of a questionnaire about the content of the visit after the preoperative visit by anesthesiology residents, including the main content of the visit, the duration of the visit, and the presumed level of patient's understanding of the anesthesia informed consent form.

Patient section:

To investigate the degree of patients' understanding of the contents of the anesthesia visit after listening to the visit. A questionnaire was used to collect the data, which included the content of the visit that the patients could recall, their level of understanding of the content explained by the physician, their concerns, and suggestions for improvement that could be taken to promote patient understanding.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Patients who have not previously undergone surgery under general anesthesia
* Patients undergoing laparoscopic cholecystectomy or laparoscopic appendectomy

Exclusion Criteria:

* Subjects who do not wish to participate in this study
* Patients with visual or auditory impairment
* Patients who are completely unable to understand the content of the communication or have communication difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age stratification of enrolled subjects, 18-80 years [young adults (18-35 years), middle-aged adults (36-60 years), older adults (61-80 years)]；
  2. Stratification of subjects' educational attainment as elementary, middle school, high school, college
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patients' understanding of the content related to anesthesia visit after the preoperative visit with anesthesiology residents | Postoperative visit （one day after surgery）
  Overall patient understanding of the anesthesia visit content was assessed by a patient self-measurement scale in the form of a rank variable, with 1 being no understanding at all and 5 being full understanding

SECONDARY OUTCOMES:
Patient recall of what anesthesiology residents mentioned during the preoperative visit vs. what anesthesiology residents mentioned during the preoperative visit | resident-side：Pre-operative visit-one day before surgery；patient-side：Post-operative visit-one day after surgery
  Differences in the content of the preoperative visit as recalled by the patient and the content of the modality as mentioned by the resident through resident-side and patient-side question and answer scales
Stratified analysis of subjects according to different age/education levels to explore the relevance in understanding the content of the preoperative visit for anesthesia | Postoperative visit （one day after surgery）
  1. Age stratification as young adults (18-35 years), middle-aged adults (36-60 years), older adults (61-80 years)；
  2. Stratification of subjects' educational attainment as elementary, middle school, high school, college.

OTHER OUTCOMES:
Patient concerns in the content of the preoperative approach | Postoperative visit （one day after surgery）
  Understanding what worries patients most about anesthesia-related content during the preoperative visit
Patients' suggestions for improving the efficiency of preoperative anesthesia visits | Postoperative visit （one day after surgery）
  Understanding what patients would like to take to promote understanding of the content of the preoperative visit from the patient's end of the spectrum

CONTACTS AND LOCATIONS:
Overall Officials: Lina Yang, Study Director
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided